CLINICAL TRIAL: NCT00782509
Title: Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 48 Weeks of Once Daily Treatment of Orally Inhaled BI 1744 CL (5 mcg [2 Actuations of 2.5 mcg] and 10 mcg [2 Actuations of 5 mcg]) Delivered by the Respimat® Inhaler, in Patients With Chronic Obstructive Pulmonary Disease (COPD
Brief Title: 12 / 48 wk Pivotal PFT vs PBO in COPD II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.12; 2008-003704-67 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

ARMS (3):
- Olodaterol (BI1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Placebo
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)

INTERVENTIONS:
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on efficacy and safety in COPD patients
  Arms: Olodaterol (BI1744) Low
Drug: Placebo — Olodaterol (BI 1744) placebo inhaled orally once daily from the Respimat inhaler
  Arms: Placebo

SUMMARY:
This primary objective of this study is to compare two doses of BI 1744 CL inhalation solution delivered by the Respimat® inhaler once daily to placebo in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion criteria:

* All patients must have a diagnosis of chronic obstructive pulmonary disease
* Male or female patients, 40 years of age or older Patients must be current or ex-smokers with a smoking history of more than 10 pack years Post bronchodilator FEV1 <80% predicted and post-bronchodilator FEV1/FVC <70%

Exclusion criteria:

* Patients with a significant disease other than COPD
* Patients with a history of asthma
* Patients with any of the following conditions:

a history of myocardial infarction within 1 year of screening visit (Visit 1) unstable or life-threatening cardiac arrhythmia. have been hospitalized for heart failure within the past year. known active tuberculosis a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed) a history of life-threatening pulmonary obstruction a history of cystic fibrosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (51):
- United States (28):
  - 1222.12.1227 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1222.12.1218 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.12.1226 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.12.1214 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1222.12.1207 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.12.1224 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1222.12.1222 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1222.12.1208 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1222.12.1220 Boehringer Ingelheim Investigational Site, River Forest, Illinois
  - 1222.12.1229 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1222.12.1219 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1222.12.1209 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1222.12.1233 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1222.12.1228 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 1222.12.1206 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1222.12.1205 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1222.12.1213 Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - 1222.12.1223 Boehringer Ingelheim Investigational Site, Harrisburg, North Carolina
  - 1222.12.1217 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1222.12.1203 Boehringer Ingelheim Investigational Site, Cincinnatti, Ohio
  - 1222.12.1201 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1222.12.1230 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1222.12.1216 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.12.1221 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1222.12.1212 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 1222.12.1211 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.12.1225 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.12.1232 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- China (11):
  - 1222.12.1298 Boehringer Ingelheim Investigational Site, Beijing
  - 1222.12.1301 Boehringer Ingelheim Investigational Site, Chongqing
  - 1222.12.1305 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1222.12.1306 Boehringer Ingelheim Investigational Site, Haikou
  - 1222.12.1302 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1222.12.1304 Boehringer Ingelheim Investigational Site, Nanjing
  - 1222.12.1296 Boehringer Ingelheim Investigational Site, Shanghai
  - 1222.12.1297 Boehringer Ingelheim Investigational Site, Shanghai
  - 1222.12.1303 Boehringer Ingelheim Investigational Site, Wuhan
  - 1222.12.1299 Boehringer Ingelheim Investigational Site, Xi'an
  - 1222.12.1300 Boehringer Ingelheim Investigational Site, Xi'an
- Germany (7):
  - 1222.12.1269 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.12.1270 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.12.1271 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.12.1268 Boehringer Ingelheim Investigational Site, Hamburg
  - 1222.12.1266 Boehringer Ingelheim Investigational Site, Koblenz
  - 1222.12.1272 Boehringer Ingelheim Investigational Site, Mannheim
  - 1222.12.1267 Boehringer Ingelheim Investigational Site, Rüdersdorf
- Taiwan (5):
  - 1222.12.1290 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1222.12.1289 Boehringer Ingelheim Investigational Site, Kaohsiung County
  - 1222.12.1288 Boehringer Ingelheim Investigational Site, Taichung
  - 1222.12.1287 Boehringer Ingelheim Investigational Site, Taipei
  - 1222.12.1286 Boehringer Ingelheim Investigational Site, Taoyuan District

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. A Post Hoc Holter ECG Analysis of Olodaterol and Formoterol in Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1955-1965. doi: 10.2147/COPD.S246353. eCollection 2020. PMID 32848381
- [Derived] Andreas S, Bothner U, Trampisch M, Haensel M, Buhl R, Alter P. Effect of long-acting beta2-agonists olodaterol and formoterol on heart rate and blood pressure in chronic obstructive pulmonary disease patients. Pulm Pharmacol Ther. 2018 Oct;52:1-6. doi: 10.1016/j.pupt.2018.08.002. Epub 2018 Aug 2. PMID 30077810
- [Derived] Ferguson GT, Feldman GJ, Hofbauer P, Hamilton A, Allen L, Korducki L, Sachs P. Efficacy and safety of olodaterol once daily delivered via Respimat(R) in patients with GOLD 2-4 COPD: results from two replicate 48-week studies. Int J Chron Obstruct Pulmon Dis. 2014 Jun 16;9:629-45. doi: 10.2147/COPD.S61717. eCollection 2014. PMID 24966672

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 644 patients were randomised into the study, however two of the patients were not treated.
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Started | 216 | 209 | 217
Completed | 175 | 185 | 181
Not Completed | 41 | 24 | 36
Not completed — Adverse Event | 20 | 10 | 20
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 5 | 8
Not completed — Non compliance with protocol | 2 | 0 | 0
Not completed — Other reasons not stated above | 5 | 2 | 3
Not completed — Lack of Efficacy | 10 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Total
Number analyzed (Participants) | 216 | 209 | 217 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.3) | 64.7 (8.1) | 65.4 (9.7) | 64.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 57 | 65 | 186
  Male | 152 | 152 | 152 | 456
Tiotropium (Tio) Use Stratum [Number; unit: Number of participants]
  Non-tiotropium | 175 | 170 | 173 | 518
  Tiotropium | 41 | 39 | 44 | 124

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first am dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose on Day 85
Population: Full analysis set (FAS). FAS is defined as all randomized patients who received at least one dose of treatment and had both baseline data and at least one post-baseline measurement at or before Day 85 (12 weeks) for either co-primary efficacy variable.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.008 (0.013) | 0.159 (0.013) | 0.152 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects model with trt,tio stratum,visit,trt-by-visit as fixed effects,baseline, baseline-by-visit as fixed covariates, patient as random effect; Mean Difference (Final Values) = 0.151, 95% CI [0.116 to 0.185], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.143, 95% CI [0.110 to 0.177], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo

2. Primary Outcome: Trough FEV1 Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h and - 10 mins prior to study drug at Day 85.
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.003 (0.014) | 0.044 (0.014) | 0.045 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.047, 95% CI [0.011 to 0.084], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0095, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.048, 95% CI [0.012 to 0.085], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-12 h (AUC 0-12h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a non-mixed effects model with treatment (trt), tio stratum, baseline as fixed effects. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and -1h and -10 min, 5 min, 15 min, 30 min, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h relative to dose at Day 85 (12 weeks)
Population: Patients in FAS with spirometry data after 3 hours at Visit 5 (12-hour pulmonary function test set)
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 98 | 116 | 107
Liter | 0.010 (0.021) | 0.120 (0.020) | 0.100 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.110, 95% CI [0.057 to 0.162], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.089, 95% CI [0.036 to 0.143], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Placebo

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline FEV1 was defined as the mean of the -1 h and -10 min measurements performed just prior to administration of the first dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit interaction as fixed categorical effects, baseline and baseline-by-visit interaction as fixed continuous covariates and patient as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose at Day 1
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Groups:
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.025 (0.013) | 0.189 (0.013) | 0.196 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.131 to 0.197], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.171, 95% CI [0.138 to 0.204], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo

5. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 2 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.025 (0.013) | 0.188 (0.013) | 0.177 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.163, 95% CI [0.130 to 0.197], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI [0.119 to 0.186], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo

6. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 6 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -1h, -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.010 (0.013) | 0.180 (0.013) | 0.171 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.135 to 0.203], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.127 to 0.195], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo

7. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 24 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | -0.010 (0.013) | 0.155 (0.013) | 0.126 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.131 to 0.200], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI [0.102 to 0.171], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

8. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve 0-3 Hour (h) (AUC 0-3h) Response After 48 Weeks
Description: as for outcome 4
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 48 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | -0.030 (0.013) | 0.132 (0.013) | 0.128 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.161, 95% CI [0.127 to 0.196], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.158, 95% CI [0.123 to 0.193], Standard Error of Mean 0.013 — Olo 10 mcg qd minus Placebo

9. Secondary Outcome: Trough FEV1 Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed a -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FEV1s if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 2 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.013 (0.014) | 0.066 (0.014) | 0.078 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0043, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.053, 95% CI [0.017 to 0.089], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.065, 95% CI [0.028 to 0.101], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

10. Secondary Outcome: Trough FEV1 Response After 6 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.002 (0.014) | 0.071 (0.014) | 0.082 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.073, 95% CI [0.037 to 0.110], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.049 to 0.121], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

11. Secondary Outcome: Trough FEV1 Response After 18 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 18 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.007 (0.014) | 0.062 (0.014) | 0.037 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [0.032 to 0.106], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.044, 95% CI [0.007 to 0.081], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

12. Secondary Outcome: Trough FEV1 Response After 24 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.036 (0.014) | 0.033 (0.014) | 0.022 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [0.032 to 0.106], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.058, 95% CI [0.021 to 0.095], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

13. Secondary Outcome: Trough FEV1 Response After 32 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 32 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.029 (0.014) | 0.029 (0.014) | -0.002 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.058, 95% CI [0.020 to 0.095], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1614, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.027, 95% CI [-0.011 to 0.064], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

14. Secondary Outcome: Trough FEV1 Response After 40 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 40 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.029 (0.014) | 0.033 (0.014) | 0.043 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.062, 95% CI [0.025 to 0.099], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.072, 95% CI [0.034 to 0.109], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

15. Secondary Outcome: Trough FEV1 Response After 48 Weeks
Description: as for outcome 2
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 48 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.057 (0.014) | 0.011 (0.014) | 0.014 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.068, 95% CI [0.031 to 0.106], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.071, 95% CI [0.033 to 0.108], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

16. Secondary Outcome: Peak FEV1 (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.099 (0.014) | 0.267 (0.014) | 0.276 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.168, 95% CI [0.132 to 0.203], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.177, 95% CI [0.142 to 0.212], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

17. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: as for outcome 16
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.104 (0.014) | 0.259 (0.014) | 0.251 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.155, 95% CI [0.119 to 0.190], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.111 to 0.182], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

18. Secondary Outcome: Peak FEV1 (0-3h) Response After 6 Weeks
Description: as for outcome 16
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 6 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.080 (0.014) | 0.252 (0.014) | 0.246 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.136 to 0.209], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.130 to 0.202], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

19. Secondary Outcome: Peak FEV1 (0-3h) Response After 12 Weeks
Description: as for outcome 16
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to -10 min, 5 min, 15 min, 30 min, 1 h, 2 h, and 3 h relative to dose after 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.088 (0.014) | 0.232 (0.014) | 0.217 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.144, 95% CI [0.108 to 0.180], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.130, 95% CI [0.094 to 0.166], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo

20. Secondary Outcome: Peak FEV1 (0-3h) Response After 24 Weeks
Description: as for outcome 16
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.062 (0.014) | 0.226 (0.014) | 0.197 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.128 to 0.201], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI [0.098 to 0.171], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

21. Secondary Outcome: Peak FEV1 (0-3h) Response After 48 Weeks
Description: as for outcome 16
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.041 (0.014) | 0.197 (0.014) | 0.198 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.155, 95% CI [0.118 to 0.192], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.157, 95% CI [0.120 to 0.194], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo

22. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hours (AUC 0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect. FVC AUC 0-3h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.052 (0.026) | 0.383 (0.026) | 0.384 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.331, 95% CI [0.263 to 0.399], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.333, 95% CI [0.265 to 0.400], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Placebo

23. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-3 Hours (AUC 0-3h) Response After 2 Weeks
Description: as for outcome 22
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.096 (0.026) | 0.338 (0.026) | 0.323 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.242, 95% CI [0.174 to 0.310], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.226, 95% CI [0.159 to 0.294], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo

24. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 6 Weeks
Description: as for outcome 22
Time Frame: as for outcome 18
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.048 (0.026) | 0.312 (0.027) | 0.294 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.263, 95% CI [0.195 to 0.332], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.246, 95% CI [0.178 to 0.315], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo

25. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 12 Weeks
Description: as for outcome 22
Time Frame: as for outcome 19
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.046 (0.026) | 0.284 (0.027) | 0.291 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.239, 95% CI [0.170 to 0.308], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.245, 95% CI [0.176 to 0.314], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo

26. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 24 Weeks
Description: as for outcome 22
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.062 (0.027) | 0.303 (0.027) | 0.281 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.241, 95% CI [0.171 to 0.311], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.219, 95% CI [0.150 to 0.289], Standard Error of Mean 0.035 — Olo 10 mcg qd minus Placebo

27. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response After 48 Weeks
Description: as for outcome 22
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.053 (0.027) | 0.271 (0.027) | 0.271 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.217, 95% CI [0.147 to 0.288], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.218, 95% CI [0.148 to 0.288], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

28. Secondary Outcome: Trough FVC Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline trough FVC was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FVC is defined as the FVCs obtained at -10 mins prior to study drug inhalation as the end of the dosing interval or the mean of -1h and -10 min FVCs if both available. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 9
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.054 (0.028) | 0.113 (0.028) | 0.141 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1040, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.059, 95% CI [-0.012 to 0.131], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0172, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.087, 95% CI [0.015 to 0.158], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

29. Secondary Outcome: Trough FVC Response After 6 Weeks
Description: as for outcome 28
Time Frame: as for outcome 10
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.029 (0.028) | 0.122 (0.028) | 0.147 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0106, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.094, 95% CI [0.022 to 0.166], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.118, 95% CI [0.046 to 0.190], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

30. Secondary Outcome: Trough FVC Response After 12 Weeks
Description: as for outcome 28
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and -1 h (if available) and - 10 mins prior to study drug after 12 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.043 (0.028) | 0.075 (0.028) | 0.091 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3821, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.032, 95% CI [-0.040 to 0.105], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1917, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.048, 95% CI [-0.024 to 0.120], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

31. Secondary Outcome: Trough FVC Response After 18 Weeks
Description: as for outcome 28
Time Frame: as for outcome 11
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.064 (0.028) | 0.114 (0.028) | 0.098 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1808, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.050, 95% CI [-0.023 to 0.123], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3700, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.033, 95% CI [-0.039 to 0.106], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

32. Secondary Outcome: Trough FVC Response After 24 Weeks
Description: as for outcome 28
Time Frame: as for outcome 12
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.021 (0.028) | 0.066 (0.028) | 0.091 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2312, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.045, 95% CI [-0.029 to 0.118], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0596, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.070, 95% CI [-0.003 to 0.144], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

33. Secondary Outcome: Trough FVC Response After 32 Weeks
Description: as for outcome 28
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.061 (0.028) | 0.099 (0.028) | 0.058 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3110, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.038, 95% CI [-0.036 to 0.111], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.9426, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.003, 95% CI [-0.076 to 0.071], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

34. Secondary Outcome: Trough FVC Response After 40 Weeks
Description: as for outcome 28
Time Frame: as for outcome 14
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | 0.062 (0.028) | 0.104 (0.028) | 0.131 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2680, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI [-0.032 to 0.115], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0662, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [-0.005 to 0.143], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

35. Secondary Outcome: Trough FVC Response After 48 Weeks
Description: as for outcome 28
Time Frame: as for outcome 15
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 205 | 205 | 207
Liter | -0.008 (0.028) | 0.038 (0.028) | 0.054 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2249, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.046, 95% CI [-0.028 to 0.120], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0994, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.062, 95% CI [-0.012 to 0.136], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

36. Secondary Outcome: FVC Peak (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Baseline FVC peak (0-3h) was defined as the mean of the available pre-dose FVC peak (0-3h) values prior to first dose of randomized treatment. FVC Peak (0-3h) values were obtained within 0 - 3 hours aftertreatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.202 (0.027) | 0.534 (0.028) | 0.535 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.332, 95% CI [0.261 to 0.403], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.333, 95% CI [0.263 to 0.403], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

37. Secondary Outcome: FVC Peak (0-3h) Response After 2 Weeks
Description: Response was defined as change from baseline. Baseline FVC peak (0-3h) was defined as the mean of the available pre-dose FVC peak (0-3h) values prior to first dose of randomized treatment. FVC Peak (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with treatment (trt), tio stratum, visit, trt-by-visit as fixed categorical effects, baseline and baseline-by-visit as fixed continuous covariates and patient as random effect.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.254 (0.027) | 0.479 (0.028) | 0.464 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.225, 95% CI [0.153 to 0.296], Standard Error of Mean 0.036 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.210, 95% CI [0.139 to 0.281], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo

38. Secondary Outcome: FVC Peak (0-3h) Response After 6 Weeks
Description: as for outcome 37
Time Frame: as for outcome 18
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.183 (0.028) | 0.451 (0.028) | 0.434 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.268, 95% CI [0.196 to 0.340], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.179 to 0.323], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

39. Secondary Outcome: FVC Peak (0-3h) Response After 12 Weeks
Description: as for outcome 37
Time Frame: as for outcome 19
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.213 (0.028) | 0.439 (0.028) | 0.422 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.226, 95% CI [0.154 to 0.298], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.209, 95% CI [0.137 to 0.281], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

40. Secondary Outcome: FVC Peak (0-3h) Response After 24 Weeks
Description: as for outcome 37
Time Frame: as for outcome 7
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.223 (0.028) | 0.449 (0.028) | 0.429 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.226, 95% CI [0.153 to 0.299], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.206, 95% CI [0.133 to 0.279], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

41. Secondary Outcome: FVC Peak (0-3h) Response After 48 Weeks
Description: as for outcome 37
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 207 | 215
Liter | 0.208 (0.028) | 0.415 (0.028) | 0.419 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI [0.133 to 0.280], Standard Error of Mean 0.037 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.211, 95% CI [0.138 to 0.285], Standard Error of Mean 0.037 — Olo 10 mcg qd minus Placebo

42. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 h (AUC 0-12h) Response at Day 85 (12 Weeks)
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Means are adjusted using a non-mixed effects model with treatment (trt), tio stratum, baseline as fixed effects. FVC AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: as for outcome 3
Population: Patients in FAS with spirometry data after 3 hours at Visit 5 (12-hour pulmonary function test set)
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 98 | 116 | 107
Liter | 0.057 (0.036) | 0.199 (0.035) | 0.212 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0028, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.142, 95% CI [0.049 to 0.235], Standard Error of Mean 0.047 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0013, ANCOVA; Treatment, tiotropium stratum and baseline as fixed effects; Mean Difference (Final Values) = 0.156, 95% CI [0.061 to 0.250], Standard Error of Mean 0.048 — Olo 10 mcg qd minus Placebo

43. Secondary Outcome: Weekly Mean Pre-dose Morning Peak Expiratory Flow Rate (PEF)
Description: Weekly mean pre-dose morning peak expiratory flow rate (PEF) at 48 weeks. PEFR measurements recorded by means of an e-Diary on a daily basis. This e-Diary was used to record the twice daily PEFs, study drug use, and rescue salbutamol (albuterol) use. The best of three readings for each measurement was recorded.
Time Frame: immediately upon arising (before drug administration) from Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 211 | 204 | 214
L/min | 182.939 (3.800) | 196.300 (3.868) | 203.873 (3.757)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0072, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 13.360, 95% CI 2-sided [3.622 to 23.099], Standard Error of Mean 4.959
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 20.934, 95% CI 2-sided [11.323 to 30.545], Standard Error of Mean 4.894

44. Secondary Outcome: Weekly Mean Evening Peak Expiratory Flow Rate (PEF)
Description: Weekly mean evening peak expiratory flow rate (PEF) at 48 weeks. PEFR measurements recorded by means of an e-Diary on a daily basis. This e-Diary was used to record the twice daily PEFs, study drug use, and rescue salbutamol (albuterol) use. The best of three readings for each measurement was recorded.
Time Frame: at bedtime from Screening to week 48
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 213 | 205 | 215
L/min | 195.502 (3.987) | 207.958 (4.065) | 216.155 (3.948)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0169, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 12.456, 95% CI 2-sided [2.242 to 22.670], Standard Error of Mean 5.201
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = 20.653, 95% CI 2-sided [10.574 to 30.731], Standard Error of Mean 5.132

45. Secondary Outcome: Weekly Mean of Daily Daytime Rescue Use
Description: The patient was to record in the e-Diary the number of puffs of salbutamol (albuterol) Metered-Dose Inhaler used each day and night. The weekly mean was calculated by taking the average of the number of puffs of rescue medication used each day during week 48.
Time Frame: Week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 205 | 215
Number of puffs | 1.363 (0.097) | 0.947 (0.099) | 0.850 (0.097)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0011, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.416, 95% CI 2-sided [-0.665 to -0.167], Standard Error of Mean 0.127
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.513, 95% CI 2-sided [-0.760 to -0.267], Standard Error of Mean 0.125

46. Secondary Outcome: Weekly Mean of Daily Nighttime Rescue Use
Description: The patient was to record in the e-Diary the number of puffs of salbutamol (albuterol) Metered-Dose Inhaler used each day and night. The weekly mean was calculated by taking the average of the number of puffs of rescue medication used each night during week 48.
Time Frame: Week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 205 | 215
Number of puffs | 2.072 (0.121) | 1.652 (0.123) | 1.312 (0.120)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0077, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.420, 95% CI 2-sided [-0.729 to -0.111], Standard Error of Mean 0.157
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.760, 95% CI [-1.065 to -0.456], Standard Error of Mean 0.155

47. Secondary Outcome: Weekly Mean of Daily (24h) Rescue Use
Description: The patient was to record in the e-Diary the number of puffs of salbutamol (albuterol) Metered-Dose Inhaler used each day and night. The weekly mean was calculated by taking the average of the number of puffs of rescue medication used each 24 hour period during week 48.
Time Frame: Week 48
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 215 | 205 | 215
Number of puffs | 3.436 (0.193) | 2.599 (0.197) | 2.158 (0.192)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0010, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -0.837, 95% CI 2-sided [-1.333 to -0.342], Standard Error of Mean 0.252
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; non-MMRM ANCOVA models with treatment, tiotropium strata and baseline as fixed effects; Mean Difference (Final Values) = -1.278, 95% CI 2-sided [-1.767 to -0.789], Standard Error of Mean 0.249

48. Secondary Outcome: Patient's Global Rating at Week 6
Description: Patients were asked to rate their respiratory condition relative to their condition prior to the first dose of study medication. The scale is a seven point scale: 1=very much better, 2=much better,3=a little better,4=no change,5=a little worse,6=much worse,7=very much worst.
Time Frame: Week 6 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 196 | 202 | 205
Point on scale | 3.3 (0.1) | 3.0 (0.1) | 2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0122, Mixed Models Analysis; Model included treatment, tiotropium stratum, visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.6 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

49. Secondary Outcome: Patient's Global Rating at Week 12
Description: as for outcome 48
Time Frame: Week 12 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 196 | 202 | 205
Point on scale | 3.2 (0.1) | 2.9 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0169, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.0], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

50. Secondary Outcome: Patient's Global Rating at Week 24
Description: as for outcome 48
Time Frame: Week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 196 | 202 | 205
Point on scale | 3.3 (0.1) | 3.0 (0.1) | 2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0180, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; [statistical method as in outcome 48, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

51. Secondary Outcome: Patient's Global Rating at Week 48
Description: as for outcome 48
Time Frame: Week 48 visit
Population: FAS
Measure: Mean (Standard Error); unit: Point on scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 196 | 202 | 205
Point on scale | 3.3 (0.1) | 3.1 (0.1) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1313, Mixed Models Analysis; Model included treatment, tiotropium stratum,visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis; Model included treatment, tiotropium stratum visit and treatment-by-visit interaction as fixed effects, patient as random; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1], Standard Error of Mean 0.1 — Olo 10 mcg qd minus Placebo

52. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor. Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank.
  The measured values presented are actually the First Quartile and 95% confidence interval.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Placebo (Tiotropium): Matching Placebo delivered by the Respimat Inhaler - tiotropium use stratum
- Placebo (Non-tiotropium): Matching Placebo delivered by the Respimat Inhaler - non-tiotropium use stratum.
- Olo 5 mcg qd (Tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 5 mcg qd (Non-tiotropium): Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
- Olo 10 mcg qd (Tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - tiotropium stratum
- Olo 10 mcg qd(Non-tiotropium): Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler - non-tiotropium stratum
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 41 | 175 | 39 | 170 | 44 | 173
days | 306.0 [98.0 to NA] — N/A indicates this statistic was not available due to the low number N/A indicates this statistic was not available due to the low number of events observed | 259.0 [169.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | 225.0 [41.0 to 336.0] | 315.0 [196.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | 219.0 [74.0 to 327.0] | 216.0 [170.0 to 307.0]
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.9853, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.993, 95% CI 2-sided [0.687 to 1.436], Standard Error of Mean 0.187 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.2344, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.241, 95% CI 2-sided [0.873 to 1.763], Standard Error of Mean 0.222 — Comparison of Olo 10 mcg qd to placebo across stratum

53. Secondary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Leading to Hospitalization
Description: Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor. Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank. The measured values presented are actually the First Quartile and 95% confidence interval.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 41 | 175 | 39 | 170 | 44 | 173
days | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [305.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [NA to NA] — N/A indicates this statistic was not available due to the low number of events observed
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.9035, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.050, 95% CI 2-sided [0.463 to 2.380], Standard Error of Mean 0.438 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.9304, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 0.958, 95% CI 2-sided [0.415 to 2.209], Standard Error of Mean 0.408 — Comparison of Olo 10 mcg qd to placebo across stratum

54. Secondary Outcome: Time to First Moderate Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Qualifying events of COPD were specifically pre-defined in the protocol.Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Moderate exacerbations were defined as exacerbations which did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids. Time to event was measured from the beginning of treatment. Cox regression analysis of treatment effect using tiotropium stratum as a stratification factor.Due to the limited number of events some statistics were not able to be calculated and are listed as N/A or are blank. The measured values presented are actually the First Quartile and 95% confidence interval..
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo (Tiotropium) | Placebo (Non-tiotropium) | Olo 5 mcg qd (Tiotropium) | Olo 5 mcg qd (Non-tiotropium) | Olo 10 mcg qd (Tiotropium) | Olo 10 mcg qd(Non-tiotropium)
Number analyzed (Participants) | 41 | 175 | 39 | 170 | 44 | 173
days | NA [211.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | 362.0 [226.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [65.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | NA [235.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | 225.0 [111.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed | 308.0 [208.0 to NA] — N/A indicates this statistic was not available due to the low number of events observed
Statistical Analysis 1: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 5 mcg qd (Tiotropium) vs Olo 5 mcg qd (Non-tiotropium); Test type: Superiority or Other; p = 0.6690, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.717 to 1.657], Standard Error of Mean 0.233 — Comparison of Olo 5 mcg qd to placebo across stratum
Statistical Analysis 2: Comparison: Placebo (Tiotropium) vs Placebo (Non-tiotropium) vs Olo 10 mcg qd (Tiotropium) vs Olo 10 mcg qd(Non-tiotropium); Test type: Superiority or Other; p = 0.1437, Log Rank; Model included a stratification factor for tiotropium use stratum and a covariate for treatment group; Hazard Ratio (HR) = 1.344, 95% CI 2-sided [0.902 to 2.002], Standard Error of Mean 0.273 — Comparison of Olo 10 mcg qd to placebo across stratum

55. Secondary Outcome: Number of COPD Exacerbations
Description: Mean number of COPD exacerbations per patient years. Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 216 | 209 | 217
COPD exacerbations | 0.4590 (0.0687) | 0.5453 (0.0765) | 0.5885 (0.0799)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3637, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.1880, 95% CI 2-sided [0.8188 to 1.7234], Standard Error of Mean 0.2251 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1853, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.2822, 95% CI 2-sided [0.8874 to 1.8527], Standard Error of Mean 0.2403 — Olo 10 mcg qd minus Placebo

56. Secondary Outcome: Number of COPD Exacerbations Requiring Hospitalization
Description: Mean number of COPD exacerbations requiring hospitalization per patient years. Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. These exacerbations required hospitalization.
Time Frame: Baseline to end of study at week 48 visit
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 216 | 209 | 217
COPD exacerbations | 0.0786 (0.0273) | 0.0811 (0.0268) | 0.0886 (0.0287)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.9455, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.0314, 95% CI 2-sided [0.4244 to 2.5063], Standard Error of Mean 0.4664 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7883, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.1273, 95% CI 2-sided [0.4696 to 2.7064], Standard Error of Mean 0.5028 — Olo 10 mcg qd minus Placebo

57. Secondary Outcome: Number of Moderate Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Mean number of moderate COPD exacerbations per patient years. Qualifying events of COPD were specifically pre-defined in the protocol. Other respiratory related events were evaluated by the investigator to see if they met the pre-defined criteria. Moderate exacerbations were defined as exacerbations which did not lead to hospitalization but included treatment with antibiotics and/or systemic steroids.
Time Frame: Baseline to end of study at 48 weeks.
Population: Treated set- all patients who received at least one dose of study medication
Measure: Mean (Standard Error); unit: COPD exacerbations
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 216 | 209 | 215
COPD exacerbations | 0.3375 (0.0587) | 0.4335 (0.0699) | 0.4513 (0.0701)
Statistical Analysis 1: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2514, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.2846, 95% CI 2-sided [0.8370 to 1.9717], Standard Error of Mean 0.2803 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1807, Negative binomial regression; Regression of treatment effect using tiotropium strata as a covariate, a log link function and log(exposure) as offset; Incidence rate ratio = 1.3373, 95% CI 2-sided [0.8735 to 2.0474], Standard Error of Mean 0.2901 — Olo 10 mcg qd minus Placebo

58. Secondary Outcome: Changes in Safety Parameters Related to Treatment
Description: Occurence of bronchoconstriction, cardiac disorders and investigations related to treatment. Bronchoconstriction is defined as any of the following events: Drop in trough FEV1 >= 15%, Rescue medication use within 30 min of inhaling randomized treatment on a clinic test day or Cough, wheeze, or dyspnoea AE within 30 min of inhaling randomized treatment on a clinic test day.
Time Frame: 48 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 216 | 209 | 217
percentage of participants
  Bronchoconstriction | 13.9 | 3.3 | 5.5
  Blood glucose increased | 0.0 | 0.5 | 0.0
  Electrocardiogram QT prolonged | 0.0 | 0.5 | 0.0
  Ventricular tachycardia | 0.0 | 1.9 | 0.5
  Ventricular extrasystoles | 0.0 | 1.0 | 1.8
  Supraventricular extrasystoles | 0.0 | 1.0 | 1.4
  Atrial fibrillation | 0.5 | 0.0 | 0.0
  Atrioventricular block | 0.0 | 0.5 | 0.0
  Atrioventricular block first degree | 0.0 | 0.5 | 0.5
  Atrioventricular block second degree | 0.0 | 0.5 | 0.0
  Bundle branch block left | 0.0 | 0.5 | 0.0
  Palpitations | 0.0 | 0.0 | 0.5
  Sinus bradycardia | 0.0 | 0.5 | 0.0
  Sinus tachycardia | 0.0 | 0.5 | 0.0

59. Secondary Outcome: Change From Baseline in Potassium
Description: Laboratory testing: Average change from baseline of potassium measured. The laboratory tests at Day 1 were considered the baseline measurements.
Time Frame: Day 1 and at 12, 24 and 48 weeks
Population: Treated set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 207 | 204 | 207
mmol/L | -0.0 (0.4) | -0.0 (0.4) | 0.0 (0.3)

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Serious Adverse Events (participants affected / at risk) | 32/216 | 32/209 | 37/217
Other Adverse Events (participants affected / at risk) | 75/216 | 71/209 | 81/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=216) | Olo 5 mcg (N=209) | Olo 10 mcg (N=217)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Lens dislocation (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3 | 5
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Aortic aneurysm (Vascular disorders) | 0 | 3 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=216) | Olo 5 mcg (N=209) | Olo 10 mcg (N=217)
Nasopharyngitis (Infections and infestations) | 18 | 19 | 25
Upper respiratory tract infection (Infections and infestations) | 17 | 20 | 22
Headache (Nervous system disorders) | 11 | 7 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 43 | 39 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication